CLINICAL TRIAL: NCT04137874
Title: Diagnostics and Triage of Acute Stroke by the National Institute of Stroke Scale (NIHSS) by Paramedics, the ParaNASPP (Paramedic - Norwegian Acute Stroke Prehospital Project) Study
Brief Title: Paramedic - Norwegian Acute Stroke Prehospital Project
Acronym: ParaNASPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Air Ambulance Foundation (Other)
Responsible Party: Principal Investigator, Maren Ranhoff Hov, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/2310
Record Dates: First submitted 2019-10-11; First posted 2019-10-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Stroke; Triage; Paramedic; Mobile Application
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: ParaNASPP is a stepped wedge cluster randomized controlled intervention trial (SW-RCT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eSTROKE (Experimental)
  Interventions: Diagnostic Test: eSTROKE model
- Control (Active Comparator): Conventional prehospital care
  Interventions: Other: Control

INTERVENTIONS:
Diagnostic Test: eSTROKE model — The eSTROKE model includes an electronic learning module, a full day course with practical teaching of National Institute of Health Stroke Scale and a mobile application which will be used for communication with in-hospital stroke physician
  Other Names: ParaNASPP
  Arms: eSTROKE
Other: Control — Conventional prehospital care
  Arms: Control

SUMMARY:
The main aim of the study is to show that patients with suspected acute stroke met by the emergency medical service and assessed using the eSTROKE model including prehospital NIHSS and a mobile application will identify a higher number of patients with stroke, than those who receive conventional prehospital care.

DETAILED DESCRIPTION:
Primary aims:

In patients with suspected stroke

1. The proportion of patients hospitalized with a suspected acute stroke and discharged with a stroke diagnose is significantly increased using the ParaNASPP model compared with conventional prehospital care
2. Time from onset to hospitalization is significantly reduced with the ParaNASPP model
3. The ParaNASPP model identifies patients eligible for direct transportation for comprehensive stroke center

ELIGIBILITY:
Inclusion Criteria:

* All patients with suspected acute stroke met by emergency medical services (ambulance and rapid response car)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Positive predictive value (PPV) of the ParaNASPP model to identify patients suffering acute stroke. | On discharge from hospital - typically within 7 days.

SECONDARY OUTCOMES:
Number of patients in hospitalized within the first 4 hours after symptom onset | first 4 hours On admission

CONTACTS AND LOCATIONS:
Locations (1):
- Prehospital services - Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fagerheim Bugge H, Guterud M, Larsen K, Toft M, Hov MR, Sandset EC. Presenting symptoms and diagnostic accuracy of prehospital stroke scales for patients with suspected mild minor stroke. Eur Stroke J. 2026 Jan 1;11(1):23969873251360592. doi: 10.1093/esj/23969873251360592. PMID 41614523
- [Derived] Fagerheim Bugge H, Guterud M, Larsen K, Toft M, Hov MR, Sandset EC. Presenting symptoms and diagnostic accuracy of prehospital stroke scales for patients with suspected mild minor stroke. Eur Stroke J. 2025 Aug 11:23969873251360592. doi: 10.1177/23969873251360592. Online ahead of print. PMID 40785620
- [Derived] Guterud M, Fagerheim Bugge H, Roislien J, Kramer-Johansen J, Toft M, Ihle-Hansen H, Bache KG, Larsen K, Braarud AC, Sandset EC, Ranhoff Hov M. Prehospital screening of acute stroke with the National Institutes of Health Stroke Scale (ParaNASPP): a stepped-wedge, cluster-randomised controlled trial. Lancet Neurol. 2023 Sep;22(9):800-811. doi: 10.1016/S1474-4422(23)00237-5. PMID 37596006
- [Derived] Bugge HF, Guterud M, Bache KCG, Braarud AC, Eriksen E, Fremstad KO, Ihle-Hansen H, Ingebretsen SH, Kramer-Johansen J, Larsen K, Roislien J, Thorsen K, Toft M, Sandset EC, Hov MR. Paramedic Norwegian Acute Stroke Prehospital Project (ParaNASPP) study protocol: a stepped wedge randomised trial of stroke screening using the National Institutes of Health Stroke Scale in the ambulance. Trials. 2022 Feb 4;23(1):113. doi: 10.1186/s13063-022-06006-4. PMID 35120559